CLINICAL TRIAL: NCT02554799
Title: A Phase 1 Exploratory Study to Evaluate the Pharmacokinetics of Selected Oral Formulations of MMV390048 Administered in the Fasted State to Healthy Volunteers
Brief Title: A Study to Evaluate the Pharmacokinetics of Oral Formulations of MMV390048 Administered Fasted to Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: Richmond Pharmacology Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: MMV_MMV390048_15_01
Record Dates: First submitted 2015-09-16; First posted 2015-09-18 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-08

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 40 mg MMV390048 tablet formulation A fasted (Experimental): 40 mg MMV390048 tablet formulation A, in fasted state
  Interventions: Drug: MMV390048 formulation A
- 40 mg MMV390048 tablet formulation B fasted (Experimental): 40 mg MMV390048 tablet formulation B fasted
  Interventions: Drug: MMV390048 formulation B
- 40 mg MMV390048 formulation A or B, with milk or fasted (Experimental): Optional cohort: 40 mg of MMV390048 in the formulation that has been shown to have the most favourable PK profile, taken with milk or in the fed state.
  Interventions: Drug: MMV390048 formulation A; Drug: MMV390048 formulation B

INTERVENTIONS:
Drug: MMV390048 formulation A — MMV390048 formulation A, tablet
  Arms: 40 mg MMV390048 formulation A or B, with milk or fasted; 40 mg MMV390048 tablet formulation A fasted
Drug: MMV390048 formulation B — MMV390048 formulation B, tablet
  Arms: 40 mg MMV390048 formulation A or B, with milk or fasted; 40 mg MMV390048 tablet formulation B fasted

SUMMARY:
This study will be conducted in a single centre, as an open single dose two parallel cohorts design with oral doses of MMV390048 administered in healthy male and female subjects between 18 to 55 years of age. Subjects will be screened within 28 days prior to entering the study. On Day 1 of the study each subject will receive one of the two MMV390048 prototype formulations, at a dose of 40 mg with 240 mL of water. Subjects will be discharged on Day 3 after 48h post-dose and they will attend the unit for follow-up visits on Days 5, 7, 10, 14, 19, 26 and 29.

DETAILED DESCRIPTION:
A Phase 1 exploratory study to evaluate the pharmacokinetics of selected oral formulations of MMV390048 administered in healthy volunteers. It is anticipated that eighteen (18) healthy male and female subjects are to be included in the study, however there is an option to include an additional cohort of 9 subjects. The optional cohort would receive a single dose of the formulation considered to have the least pharmacokinetic variability with a suitable safety and tolerability profile with food or milk. Timing of PK samples may be adjusted in accordance with evolving data and dosing schedule. Additional or fewer PK samples may be taken in accordance with evolving data and dosing schedule to establish full protocol specific PK profile. The study specific maximum blood volume taken will not be exceeded.

ELIGIBILITY:
Inclusion Criteria:

* healthy male or female (non-childbearing potential) of any race, aged 18 to 55 years
* body weight at least 50kg and a body mass index 18 to 30Kg/m2
* Females must be of non-childbearing potential:

  * Natural (spontaneous) post-menopausal defined (amenorrheic for at least 12 months without an alternative medical cause with a screening follicle stimulating hormone level >25IU/L (for post-menopause).
  * Premenopausal with irreversible surgical sterilization by hysterectomy
  * and/or bilateral oophorectomy or salpingectomy at least 6 months before screening
* Males agree to use acceptable methods of contraception if the male subject's partner could become pregnant from the time of study medication until 120 days after administration of study medication. One of the following acceptable methods of contraception must be used:

  * Condom and occlusive cap (diaphragm or cervical/vault cap) with spermicidal foam/gel/film/cream/suppository
  * Surgical sterilization (vasectomy with documentation of azoospermia) and an acceptable barrier method (condom or occlusive cap [diaphragm or cervical/vault cap] used with spermicidal foam/gel/film/cream/suppository)
  * subject's female partner uses oral contraceptives (combination estrogen / progesterone pills), injectable progesterone or sub-dermal implants and an acceptable barrier method
  * subject's female partner uses medically prescribed topically applied transdermal contraceptive patch and an acceptable barrier method
  * subject's female partner has undergone documented tubal ligation (female sterilization). In addition, an acceptable barrier method must be used.
  * subject's female partner has undergone documented placement of an intrauterine device or intrauterine system. In addition, an acceptable barrier method must be used.
  * True abstinence: when in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception. Abstinent subjects have to agree to use 1 of the above-mentioned contraceptive methods, if they start sexual relationships during the study and for up to 120 days post-study drug
* non-smokers or ex-smokers for more than 90 days prior to screening or smoke no more than 5 cigarettes per day. If users of nicotine products (spray, patch, e-cigarette, etc.) they should use the equivalent of no more than 5 cigarettes /day
* Subjects should not donate egg or sperm from the time of administration of study medication until 120 days post-study drug
* capable of fully understanding and complying with the requirements of the study and must sign the informed consent form prior to undergoing any study-related procedures
* agree to avoid excessive UV radiation exposure (occupational exposure to the sun, sunbathing, tanning salon use, phototherapy, etc.) throughout the study.

Exclusion Criteria:

* Male subjects with a female partner(s) who is (are) pregnant or lactating from the time of study medication
* Women of childbearing potential, defined as all women physiologically capable of becoming pregnant, including women whose career, lifestyle, or sexual orientation precludes intercourse with a male partner and women whose partners have been sterilized by vasectomy or other means
* Current or recurrent disease (e.g. cardiovascular, neurological, renal, gastrointestinal, oncologic or other conditions) that may affect the action, absorption or disposition of the study medication or could affect clinical assessments or clinical laboratory evaluations
* Current or relevant history of physical or psychiatric illness that may require treatment or make the subject unlikely to fully comply with the requirements or complete the study, or any condition that presents undue risk from the investigational product or study procedures
* Any other significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk because of the participation in the study, may influence the result of the study, or the subject's ability to participate in the study
* History of photosensitivity
* History or clinical evidence of alcohol or substance abuse. Alcohol abuse is defined as regular weekly intake of more than 21 units for males and 14 units for females
* Any clinically relevant history of intolerance/allergy to milk or dairy products
* Use of an investigational product or participation in a clinical study within 90 days before study medication
* Donation of blood products or of more than 500ml of blood in 90 days prior to study medication
* Use of any prescription drugs within 14 days or within 5 times the elimination half-life (whichever period is longer) prior to study medication
* Use moderate or strong inhibitors and/or inducers of CYP450/Transporters within 4 weeks prior to study drug administration (or 5 half-lives of the compound if longer)
* Use of over-the-counter medications or dietary supplements, including vitamins and herbal supplements within 7 days of study drug. With the exception of paracetamol which may be used incidentally or for short-term treatment at a maximum of 2g/day
* Intake of grapefruit, grapefruit juice or other products containing grapefruit within 28 days prior to study drug
* Excessive intake of caffeine drinks or energy drinks within 48 hours before admission (more than three 250ml cups of coffee a day, equivalent to roughly 250mg caffeine)
* Any clinically significant abnormal laboratory, vital signs or other safety findings as determined by medical history, physical examination or other evaluations at screening or admission.
* Any liver function tests elevated >1.5 times the upper limit of normal, considered by the investigator as clinically relevant, at screening or admission
* Abnormal serum Hemoglobin, Haptoglobin, Reticulocyte count or Lactate Dehydrogenase at screening/admission
* abnormal ECG results at screening/admission results considered as clinically significant by the investigator
* Confirmed positive urine drug screen (amphetamines, benzodiazepines, cocaine, cannabinoids, opiates, barbiturates or methadone) or from the alcohol breath test at screening/admission.
* positive human immunodeficiency virus, hepatitis B surface antigen, anti Hepatitis core antibody, or hepatitis C virus antibody at screening
* veins unsuitable for intravenous puncture or cannulation on either arm (e.g. veins difficult to locate, access or puncture, veins with a tendency to rupture during or after puncture) 23. Any conditions which in the opinion of the investigator would make the subject unsuitable for enrolment or could interfere with the subjects' participation in or completion of the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-09-17 (Actual); Primary Completion 2015-10-28 (Actual); Study Completion 2015-10-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Richmond Pharmacology Ltd., Croydon, London, United Kingdom

REFERENCES:
- [Derived] Sinxadi P, Donini C, Johnstone H, Langdon G, Wiesner L, Allen E, Duparc S, Chalon S, McCarthy JS, Lorch U, Chibale K, Mohrle J, Barnes KI. Safety, Tolerability, Pharmacokinetics, and Antimalarial Activity of the Novel Plasmodium Phosphatidylinositol 4-Kinase Inhibitor MMV390048 in Healthy Volunteers. Antimicrob Agents Chemother. 2020 Mar 24;64(4):e01896-19. doi: 10.1128/AAC.01896-19. Print 2020 Mar 24. PMID 31932368

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Optional Cohort:
  The study design of this clinical trial allowed for an optional cohort to be enrolled. Ultimately, such optional cohort was not deemed required and therefore not conducted.
Groups:
- 40 mg MMV390048 Form A Fasted: 40 mg MMV390048 tablet formulation A fasted
- 40 mg MMV390048 Form B Fasted: 40 mg MMV390048 tablet formulation B fasted
Period: Overall Study
Arm/Group | 40 mg MMV390048 Form A Fasted | 40 mg MMV390048 Form B Fasted
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 40 mg MMV390048 Form A Fasted | 40 mg MMV390048 Form B Fasted | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Continuous [Median (Standard Deviation); unit: years] | 29 (10.37) | 26 (11.5) | 28.5 (10.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 9 | 9 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 9 | 8 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 5 | 7 | 12
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Cmax: Peak Plasma Concentration
Description: Maximum concentration (Cmax) of two MMV390048 prototype formulations administered in the fasted state
Time Frame: Up to 672 hours post-dose
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 40 mg MMV390048 Form A Fasted | 40 mg MMV390048 Form B Fasted
Number analyzed (Participants) | 9 | 9
ng/mL | 277 (62.5) | 373.4444 (64.7825)

2. Primary Outcome: Tmax: Time to Reach Peak Plasma Concentration
Description: Time to reach maximum plasma concentration (Tmax) of two MMV390048 prototype formulations administered in the fasted state
Time Frame: Up to 672 hours post-dose
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 40 mg MMV390048 Form A Fasted | 40 mg MMV390048 Form B Fasted
Number analyzed (Participants) | 9 | 9
hours | 2.4 (1.01) | 2.6 (0.53)

3. Primary Outcome: AUC: Area Under the Plasma Concentration-time Curve From Zero to Infinity
Description: Area under the plasma concentration-time curve (AUC) of two MMV390048 prototype formulations administered in the fasted state
Time Frame: From Pre-dose to 672 hours post-dose
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | 40 mg MMV390048 Form A Fasted | 40 mg MMV390048 Form B Fasted
Number analyzed (Participants) | 9 | 9
h*ng/mL | 56991.64 (39197.535) | 63228.3 (29689.434)

4. Primary Outcome: Terminal Elimination Half-life (t1/2)
Description: Terminal elimination half-life (t1/2) of two MMV390048 prototype formulations administered in the fasted state
Time Frame: Up to 672 hours post-dose
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 40 mg MMV390048 Form A Fasted | 40 mg MMV390048 Form B Fasted
Number analyzed (Participants) | 9 | 9
hours | 192.0663 (90.5336) | 160.3984 (61.3228)

5. Primary Outcome: Terminal Elimination Rate Constant (Lambda z)
Description: Terminal elimination rate constant (lambda z) of two MMV390048 prototype formulations administered in the fasted state
Time Frame: Up to 672 hours post-dose
Measure: Mean (Standard Deviation); unit: 1/hours
Arm/Group | 40 mg MMV390048 Form A Fasted | 40 mg MMV390048 Form B Fasted
Number analyzed (Participants) | 9 | 9
1/hours | 0.0041 (0.0011) | 0.0051 (0.0024)

6. Primary Outcome: Oral Plasma Clearance (CL/F)
Description: Oral plasma clearance (CL/F) of two MMV390048 prototype formulations administered in the fasted state
Time Frame: Up to 672 hours post-dose
Measure: Mean (Standard Deviation); unit: L/hours
Arm/Group | 40 mg MMV390048 Form A Fasted | 40 mg MMV390048 Form B Fasted
Number analyzed (Participants) | 9 | 9
L/hours | 0.8819 (0.3473) | 0.7635 (0.3658)

7. Primary Outcome: Apparent Volume of Distribution (Vz/F)
Description: Apparent volume of distribution (Vz/F) of two MMV390048 prototype formulations administered in the fasted state
Time Frame: Up to 672 hours post-dose
Measure: Mean (Standard Deviation); unit: Litres
Arm/Group | 40 mg MMV390048 Form A Fasted | 40 mg MMV390048 Form B Fasted
Number analyzed (Participants) | 9 | 9
Litres | 211.9523 (45.8906) | 155.3750 (49.9488)

8. Other Pre Specified Outcome: Time to Reach Maximum Plasma Concentration (Tmax)
Description: Exploratory: Time to reach maximum plasma concentration of one MMV390048 prototype formulation administered with food or milk
Time Frame: Up to 672 hours post-dose
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Area Under the Plasma Concentration-time Curve (AUC)
Description: Exploratory: Area under the plasma concentration-time curve from zero to infinity of one MMV390048 prototype formulation administered with food or milk
Time Frame: Up to 672 hours post-dose
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Terminal Elimination Half-life
Description: Exploratory: Terminal elimination half-life of one MMV390048 prototype formulation administered with food or milk
Time Frame: Up to 672 hours post-dose
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Terminal Elimination Rate Constant
Description: Exploratory: terminal elimination rate constant of one MMV390048 prototype formulation administered with food or milk
Time Frame: Up to 672 hours post-dose
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Oral Plasma Clearance
Description: Exploratory: Oral plasma clearance of one MMV390048 prototype formulation administered with food or milk
Time Frame: Up to 672 hours post-dose
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Apparent Volume of Distribution
Description: Exploratory: Apparent volume of distribution of one MMV390048 prototype formulation administered with food or milk
Time Frame: Up to 672 hours post-dose
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 672 hours post-dose (=study completion)
Arm/Group | 40 mg MMV390048 Form A Fasted | 40 mg MMV390048 Form B Fasted
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 4/9 | 3/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 40 mg MMV390048 Form A Fasted (N=9) | 40 mg MMV390048 Form B Fasted (N=9)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 2 (2) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament Sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Richmond Pharmacology Limited (RPL) shall not issue or submit any press release for publication without MMV's prior written approval.

In recognition that RPL and the Site Principal Investigator have a responsibility to ensure that results of scientific interest arising from a Clinical Trial are appropriately published and disseminated, RPL may, upon MMV's written consent which will not be unreasonably withheld, publish Results of a clinical trial carried out under a Project Agreement.